CLINICAL TRIAL: NCT03986203
Title: Evaluation of the Spry Belt for Improving Bone Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theranova, L.L.C. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRD-09-1257; R44AG046005 (NIH)
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Osteopenia
Keywords: Low bone mass; Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the clinical site staff member who trains the subject will know the group assignment. All subsequent interactions with each subject will not be carried out by the trainer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active (Experimental): Subjects in this group will receive the active treatment for each daily treatment session.
  Interventions: Device: Spry Belt
- Sham (Sham Comparator): Subjects in this group will receive the sham treatment for each daily treatment session.
  Interventions: Device: Spry Belt

INTERVENTIONS:
Device: Spry Belt — The Spry Belt delivers energy to the user that may help prevent bone loss. Participants will wear the device for 30 minutes a day, 5 days a week for one year. The active and sham devices are identical except for the specific energy that is delivered to the user.

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of the Spry Belt. The Spry Belt is intended to deliver energy to the user's skeleton to reduce the progression of age-related decrease in bone quality in postmenopausal women. Half of the participants will receive the active treatment, while the other half will receive the sham/placebo treatment.

DETAILED DESCRIPTION:
Women lose a significant amount of bone after menopause and are at high risk of breaking bones. Bone cells have been shown to be responsive to different forms of applied energy, which can be used to reduce the progression of age-related declines in bone properties. The purpose of this research study is to evaluate the safety and effectiveness of the Spry Belt when used regularly over one year. The Spry Belt, a medical device that is worn around the hips like a belt, provides energy to the user's skeleton with the goal of improving bone quality in postmenopausal women with osteopenia, or low bone mass.

In this randomized, controlled study, all participants will receive the Spry Belt for at-home use over the 12 month study. Participants will be randomized (1:1) to the active or sham/placebo treatment group and give a Spry Belt that is pre-programmed to deliver the corresponding therapy. Participants will self-administer treatment sessions at least 5 times per week for 12 months. The effectiveness of the Spry Belt treatment will be assessed via CT and DXA scans of the user's bones to evaluate changes in bone density and strength over the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Had her last menstrual period at least one year prior to the time of study enrollment
* Has low bone mass as defined by a DXA T-score between -1.0 and -2.49 for the femoral neck, proximal femur, total femur, or lumbar spine
* Is 50 years of age or older
* Can walk and stand without an assistive device
* Is able to provide informed consent
* Is able to understand spoken and written English
* Is capable and willing to follow all study-related procedures

Exclusion Criteria:

* Has a bone mineral density (BMD) at the femoral neck, proximal femur, total femur, or lumbar spine of T score ≤ -2.5 (defined by DXA)
* Has a 10-year probability of major fracture >20% or hip fracture >3% based on results of the Fracture Risk Assessment (FRAX) Tool
* Is currently taking or has taken bisphosphonates or other prescription osteoporosis medications in the past 24 months, or estrogen replacement therapy, glucocorticosteroids, or other drugs affecting bone in the past 3 months
* Has had at least one fracture or at least one major surgery within the past 6 months
* Smokes >10 cigarettes per day over the past 6 months
* Has had an average of 14 alcoholic drinks per week over the past 6 months
* Has type I diabetes
* Has a history of severe renal disease or kidney failure
* Has had gastric bypass surgery
* Has been diagnosed with chronic renal disease, cirrhosis, multiple myeloma, neuromuscular disease, osteomalacia, Paget's disease, osteogenesis imperfecta, severe osteoarthritis, rheumatoid arthritis, severe peripheral neuropathy, gastrointestinal malabsorption or sprue, an eating disorder (e.g., anorexia nervosa, bulimia), uncontrolled hypertension, or chronic diseases known to affect the musculoskeletal system (e.g., muscular dystrophy)
* Has been diagnosed with an endocrine disorder known to adversely affect bone density, such as hyperparathyroidism, hyperthyroidism, or Cushing's syndrome
* Has cancer and/or is being treated for cancer
* Has had a bilateral oophorectomy
* Is being treated for a herniated disc
* Has had any prolonged immobilization (i.e., bedrest) for over one week or non-weight bearing for greater than one month of the axial or lower appendicular skeleton within the last 3 years
* Is engaged in high-impact activity at least three times per week (including but not limited to tennis, aerobics, running, weight-bearing activity or exercise more intense than fast walking).
* Has a known allergy to neoprene
* Has a hip circumference >56 inches
* Has a BMI > 35
* Has abnormal results for the following laboratory tests:

  * Serum 25(OH)D outside of the range: 10-100 ng/mL
  * Serum calcium outside of the range: 8.9-10.3 mg/dL
  * Serum PTH outside of the range: 12-88 pg/mL
  * TSH outside of the range: 0.4 - 5.0 mIU/L (Note: If lab results are abnormal, subjects may see their MD to have thyroid medication adjusted and may be re-screened. If results are within the normal range, they may proceed with enrollment.)
  * FSH less than 40 (mIU/L) (Note: FSH will be analyzed to confirm menopause, when necessary, such as in cases where women have had a history of hysterectomy and unilateral oophorectomy.)
* Has joint replacement implants in the ankle, knee, or hip
* Has had a spinal fusion procedure
* Has an active implant (e.g. implanted neurostimulator) in the areas of the lumbar or thoracic spine, pelvis, or buttocks
* Has had a major change in high-impact physical activity level (increase or decrease) in the past 3 months
* Has undergone or is undergoing transgender hormone therapy
* Is deemed unsuitable for enrollment in the study by the Principal Investigator

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-08-13 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Vertebral body strength | Change from baseline to 12 months
  Change in lumbar vertebral body strength as estimated via finite element analysis from CT scan data. A higher value indicates higher strength.
Number of device-related adverse events present | 12 months
  Safety assessment via device-related adverse events

SECONDARY OUTCOMES:
Vertebral body bone mineral density | Change from baseline to 12 months
  Change in lumber vertebral body areal bone mineral density (BMD) as assessed via dual-energy x-ray absorptiometry (DXA) scan. A higher BMD value indicates higher bone density.
Femoral bone mineral density | Change from baseline to 12 months
  Change in femoral areal bone mineral density (BMD) as assessed via dual-energy x-ray absorptiometry (DXA) scan. A higher BMD value indicates higher bone density.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bilek, PT, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No